CLINICAL TRIAL: NCT00225264
Title: A Double-Blind, Randomized, Comparator-Controlled Study in Subjects With Type 2 Diabetes Mellitus Comparing the Effects of Pioglitazone HCl Versus Glimepiride on the Rate of Progression of Atherosclerotic Disease as Measured by Carotid Intima-Media Thickness
Brief Title: Efficacy Study of Pioglitazone and Glimepiride on the Rate of Progression of Atherosclerotic Disease.
Acronym: CHICAGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-02-TL-OPI-518; U1111-1114-2799 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone QD (Experimental)
  Interventions: Drug: Pioglitazone
- Glimepiride QD (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 15 mg titrated up to 45 mg, tablets, orally, once daily and glimepiride placebo-matching capsules, orally, once daily for up to 72 weeks.
  Other Names: Actos; AD-4833
  Arms: Pioglitazone QD
Drug: Glimepiride — Pioglitazone placebo-matching tablets, orally, once daily and glimepiride 1 mg titrated up to 4 mg, capsules, orally, once daily for up to 72 weeks.
  Other Names: Amaryl
  Arms: Glimepiride QD

SUMMARY:
The primary purpose of this study is to compare the effects of pioglitazone, once daily (QD), versus glimepiride on the amount of thickening of the carotid artery.

DETAILED DESCRIPTION:
Diabetes is a chronic disease with multiple metabolic defects that result in hyperglycemia arising from inadequate insulin activity. Type 2 diabetes usually is the result of a progression from reduced sensitivity of hepatic and peripheral tissue cells to circulating insulin to a progressive inability of the body to produce adequate insulin to overcome insulin resistance, resulting in impaired glucose tolerance and ultimately overt diabetes. In the United States, an estimated 21 million people have diabetes, with type 2 diabetes occurring in approximately 90% to 95% of cases.

Type 2 diabetes also represents an important risk group for the development of accelerated atherosclerosis. Atherosclerosis can be measured with different procedures. One of the noninvasive, commonly used procedures is carotid B-mode ultrasound measurement of carotid intima-media thickness, which has been shown to be a useful measurement for clinical cardiovascular events in multiple studies.

Coronary artery calcification is a marker of coronary artery disease, and electron beam tomography is a sensitive tool for evaluation of coronary artery calcium. Electron beam tomography measurements produce a coronary artery calcium score that represents plaque burden. Subjects with diabetes mellitus have accelerated coronary artery disease. Even after treatment of elevated lipid levels, rates for coronary events still exceed those seen in non-diabetic subjects treated with the same lipid-lowering agents. Diabetic subjects also continue to have increased mortality rates compared with non-diabetic subjects after a myocardial infarction. Therefore, detection of sub-clinical atherosclerosis and prevention of myocardial infarction in subjects with diabetes remains an important priority.

Pioglitazone is a thiazolidinedione developed by Takeda Chemical Industries, Ltd, and depends on the presence of insulin for its mechanism of action. Data suggests that thiazolidinediones may inhibit the development of atherosclerosis in non-diabetic, atherosclerosis mouse models. These findings suggest that this class of drugs may have an effect on vessel walls to suppress development of atherosclerotic lesions.

This study will investigate the effects of pioglitazone and glimepiride on the rate of progression of atherosclerotic disease as measured by carotid intima-media thickness and by electron beam tomography of the coronary arteries in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study. Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to the time of randomization.
* Diagnosis of type 2 diabetes mellitus.
* Has received appropriate counseling on lifestyle modification for type 2 diabetes, including diet and exercise.
* Naïve to or not currently taking antidiabetic therapy, or is currently treated with monotherapy or combination antidiabetic therapy.
* Glycosylated hemoglobin greater than or equal to 6.0% and less than 9% at screening if taking antidiabetic medication or glycosylated hemoglobin greater than or equal to 6.5% and less than 10% at screening if naïve to or not taking antidiabetic medication.

Exclusion Criteria

* Type 1 diabetes mellitus.
* Taking more than 2 antidiabetic therapies at screening. For combination medications, each component is counted as 1 therapy.
* Symptomatic coronary artery disease, cerebrovascular disease, or peripheral vascular disease at the time of screening.
* Taking or have taken pioglitazone or other thiazolidinediones within 12 weeks of randomization or were discontinued from thiazolidinedione therapy due to lack of efficacy or clinical or laboratory signs of intolerance.
* Was discontinued from glimepiride or other sulfonylureas due to lack of efficacy or clinical or laboratory signs of intolerance.
* Participating in another investigational study or has participated in an investigational study within the past 30 days or is scheduled to participate in an investigational study during the time frame of this study.
* Women who are pregnant, intend to become pregnant during the course of the study, or are lactating.
* Men who have serum creatinine greater than or equal to 2.0 mg/dL (greater than or equal to 1.5 mg/dL if taking metformin) and women with serum creatinine greater than or equal to 1.8 mg/dL (greater than or equal to1.4 mg/dL if taking metformin).
* Unexplained microscopic hematuria of greater than plus 1 confirmed by repeat testing.
* History of drug abuse or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 2 years.
* Clinical cardiac failure as defined by New York Heart Association class III or IV, or known left ventricular dysfunction measured as left ventricular ejection fraction less than 40%, or by current use of diuretics or angiotensin converting enzyme inhibitors for the treatment of heart failure. Use of these agents for other therapeutic reasons is not an exclusion.
* Alanine transaminase level of greater than 2.5 times the upper limit of normal, active liver disease or jaundice.
* Weighs greater than 300 pounds or has a body mass index greater than 45 kg/m2 as calculated by weight (kg)/height (m)2 or weight (pounds)/height (inches)2 x 703.
* Has taken excluded medications.
* Known or suspected malignancy or recurrence of malignancy within the past 5 years, with the exception of basal cell carcinoma and Stage 1 squamous cell carcinoma of the skin.
* Any disease where, in the opinion of the investigator, survival is expected to be less than 18 months.
* Anticipated to undergo coronary bypass surgery or cardiac intervention during the course of the study.
* Has, in the opinion of the investigator, clinically significant valvular heart disease likely to require surgical repair or replacement during the course of the study.
* Has had uncontrolled hypertension (ie, sitting systolic blood pressure greater than160 mm Hg or sitting diastolic blood pressure greater than 100 mm Hg) at randomization.
* Men who have hemoglobin less than10.5 g/dL and women who have hemoglobin less than10.0 g/dL.
* Triglycerides greater than 500 mg/dL.
* Unwilling or unable to comply with the protocol or scheduled appointments.
* Unable to understand verbal and/or written English or any other language for which a certified translation of the informed consent is available.
* Known or suspected hypersensitivity to blood, blood products, or albumin.
* Subjects for whom it is not possible to obtain good quality images of the common carotid artery for technical reasons.
* Potentially clinically significant stenosis of the carotid artery as determined according to current guidelines by the physician assessing carotid intima-media thickness results. In these cases, the carotid intima-media thickness results should be reviewed by the investigator in consultation with the carotid intima-media thickness physician prior to determining whether the subject should be randomized.
* Has had bilateral endarterectomies, bilateral carotid stents, or radiation to the head or neck.
* Has received radiation therapy in the past year, who has had more than one computed tomography scan in the past year, or who is unable to raise one's arms above one's head while in a prone position.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2003-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Absolute change from Baseline in carotid intima-media thickness. | Weeks 24, 48 and Final Visit.

SECONDARY OUTCOMES:
Change from Baseline in carotid intima-media thickness. | Weeks 24, 48 and Final Visit.
Change from Baseline in coronary artery calcium-volume score. | At Final Visit
Change from Baseline in abdominal adipose tissue content and distribution. | At Final Visit
Incidence of cardiovascular events as a composite of cardiovascular mortality, nonfatal myocardial infarction and nonfatal stroke | At each occurrence
Incidence of cardiovascular events as a composite of cardiovascular mortality, nonfatal MI, nonfatal stroke, coronary revascularization, carotid endarterectomy/stenting, hospitalization for unstable angina and hospitalization for CHF | At each occurrence

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (1):
- Chicago, Illinois, United States

REFERENCES:
- [Result] Mazzone T, Meyer PM, Feinstein SB, Davidson MH, Kondos GT, D'Agostino RB Sr, Perez A, Provost JC, Haffner SM. Effect of pioglitazone compared with glimepiride on carotid intima-media thickness in type 2 diabetes: a randomized trial. JAMA. 2006 Dec 6;296(21):2572-81. doi: 10.1001/jama.296.21.joc60158. Epub 2006 Nov 13. PMID 17101640
- [Result] Davidson M, Meyer PM, Haffner S, Feinstein S, D'Agostino R Sr, Kondos GT, Perez A, Chen Z, Mazzone T. Increased high-density lipoprotein cholesterol predicts the pioglitazone-mediated reduction of carotid intima-media thickness progression in patients with type 2 diabetes mellitus. Circulation. 2008 Apr 22;117(16):2123-30. doi: 10.1161/CIRCULATIONAHA.107.746610. Epub 2008 Apr 14. PMID 18413496
- [Result] Sam S, Haffner S, Davidson MH, D'Agostino RB Sr, Feinstein S, Kondos G, Perez A, Mazzone T. Relationship of abdominal visceral and subcutaneous adipose tissue with lipoprotein particle number and size in type 2 diabetes. Diabetes. 2008 Aug;57(8):2022-7. doi: 10.2337/db08-0157. Epub 2008 May 9. PMID 18469202
- [Result] Mazzone T, Meyer PM, Kondos GT, Davidson MH, Feinstein SB, D'Agostino RB Sr, Perez A, Haffner SM. Relationship of traditional and nontraditional cardiovascular risk factors to coronary artery calcium in type 2 diabetes. Diabetes. 2007 Mar;56(3):849-55. doi: 10.2337/db06-0935. PMID 17327456
- [Result] Sam S, Haffner S, Davidson MH, D'Agostino RB Sr, Feinstein S, Kondos G, Perez A, Mazzone T. Relation of abdominal fat depots to systemic markers of inflammation in type 2 diabetes. Diabetes Care. 2009 May;32(5):932-7. doi: 10.2337/dc08-1856. Epub 2009 Feb 19. PMID 19228869
- [Result] Betteridge DJ. CHICAGO, PERISCOPE and PROactive: CV risk modification in diabetes with pioglitazone. Fundam Clin Pharmacol. 2009 Dec;23(6):675-9. doi: 10.1111/j.1472-8206.2009.00741.x. Epub 2009 Sep 10. PMID 19744248
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI